CLINICAL TRIAL: NCT02997358
Title: Randomised Phase III Multicentric Study Comparing Efficacy of Doxorubicin With Trabectedin Followed by Trabectedin in Non-progressive Patients Versus Doxorubicine Alone as First-line Therapy in Patients With Metastatic or Unresectable Leiomyosarcoma (Uterine or Soft Tissue)
Brief Title: Study Comparing Efficacy of Doxorubicin With Trabectedin Followed by Trabectedin Versus Doxorubicine in Patients With Leiomyosarcoma
Acronym: LMS04
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-002186-56; 2016/2410 (Other: CSET number)
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Uterine or Soft Tissue Leiomyosarcoma
MeSH Terms: interventions — Doxorubicin; Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxorubicin (Active Comparator): 6 cycles - 1 cycle every 3 weeks (day 1 to day 21) On day 1: Doxorubicin 75 mg/m² IV
  Interventions: Drug: Doxorubicin
- doxorubicin + trabectedin followed by maintenance trabectedin (Experimental): 1. Doxorubicin + trabectedin 6 cycles - 1 cycle every 3 weeks (day 1 to day 21) Doxorubicin 60 mg/m² IV D1, then Trabectedin 1.1 mg/m² per CIV 3 hours D1. Surgery for residual disease is possible after 6 cycles (in case of non evolutive disease)
  2. In case of response or stable disease after 6 cycles 3-weeks cycle until disease progression or for a maximum of 12 months of treatment (maximum 17 cycles in maintenance therapy), whichever occurs first Trabectedin 1.1 mg/m² per CIV 3 hours
  Interventions: Drug: Doxorubicin; Drug: Trabectedin

INTERVENTIONS:
Drug: Doxorubicin — 75 mg/m² Day 1 of each 3-weeks cycle
Drug: Trabectedin — 150 μg/m²/day s.c From day 3 to day 9
  Arms: doxorubicin + trabectedin followed by maintenance trabectedin

SUMMARY:
The objective of LMS04 study is to better define the treatment strategy for patients with metastatic leiomyosarcoma (uterine or soft tissue), as well as identifying the best first line therapeutic option for these patients. LMS04 will test a new strategy for first line therapy LMS sarcoma compare to the reference therapy (6 cycles of doxorubicin alone): the interest of the association of trabectedin to doxorubicin in first line treatment followed by trabectedin alone for non-progressive patients after 6 cycles of the association of trabectedin and doxorubicin (the LMS02 design).

LMS04 will be the first phase III randomized study specifically dedicated to soft tissue leiomyosarcoma in first line metastatic disease.

It is planned to compare a new doxorubicin combination (including trabectedin) with very encouraging results followed by trabectedin maintenance therapy for non-progressive patients to doxorubicin alone. Prospective ancillary translational studies will attempt to define profiles of patients who could benefit from this new chemotherapy in an exploratory way.

The validation of a new first line option specific for LMS, identifying clinical factors that characterize aggressiveness and responsiveness to treatment aims to have an important in the spirit of personalized medicine in this rare and deadly disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed diagnosis of metastatic or relapsed unresectable uterine or soft tissue leiomyosarcoma, reviewed in a reference center (among RREPS network), previously untreated with chemotherapy , and with available Formalin Fixed Paraffin Embedded (FFPE) blocks
2. At least one measurable lesion according to RECIST V 1.1 criteria. Target could be in a previously irradiated field but has to be progressive or a biopsy had to be positive before inclusion.
3. Age ≥ 18 years old
4. ECOG performance status < 2 (Appendix 4)
5. Adequate haematological, liver and cardiac functions:

   * Neutrophil counts ≥ 1500/mm3
   * Platelets ≥ 100 000/mm3
   * Serum creatinin < 1.5 x Upper Limit of Normal Value (UNL)
   * Serum bilirubin ≤1 x ULN
   * ALT, AST ≤ 2.5 x ULN
   * Alcaline phosphatases ≤ 1.5 x ULN
   * Cardiac ultrasound and/or normal isotopic ventriculography : Shortening Fraction (SF) > 30%, Left Ventricular Ejection Fraction (LVEF) > 50%
6. Creatinin phosphokinase (CPK) ≤ 2.5 x ULN
7. Women of childbearing potential (WOCBP) must have a negative pregnancy test within 7 days prior to inclusion. Both males and WOCBP who are sexually active should be using an effective birth control method from inclusion (for WOCBP) or treatment initiation (for male) and up to 6 months following the last dose of study drug.
8. Signed written informed consent form
9. Patient affiliated to a social security regimen or beneficiary of the same

Exclusion Criteria:

1. All other histological types of uterine sarcomas or soft tissue sarcomas
2. Any contraindication for the use of trabectedin and/or doxorubicin (cardiac, renal, hepatic, known hypersensitivity…)
3. Patient already enrolled in another therapeutic trial involving an investigational substance, and when such a substance has been taken during the previous 4 weeks.
4. Medical history of progressive psychiatric disorder
5. History of another type of cancer not in complete remission for more than 3 years prior to study entry (except for cutaneous basal cell carcinoma or in situ cervical epithelioma), and/or having required any chemotherapy treatment at any time.
6. Known cerebral metastasis
7. History of allograft or autograft
8. Active viral hepatitis B or C or known human immunodeficiency virus (HIV) infection or any other uncontrolled infection
9. Pregnant women or nursing mothers
10. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or any condition (e.g., psychological instability, geographical location, social reason, etc.) that, in the judgment of the Investigator, may affect the patient's ability to understand and sign the informed consent or to fully comply with all study visits, treatments, procedures, and other requirements scheduled in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Progression free Survival | Until progression or 2 years after randomization, whichever occurs first
  Tumour assessment will be analysed using RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pautier P, Italiano A, Piperno-Neumann S, Chevreau C, Penel N, Firmin N, Boudou-Rouquette P, Bertucci F, Lebrun-Ly V, Ray-Coquard I, Kalbacher E, Bompas E, Collard O, Isambert N, Guillemet C, Rios M, Le Cesne A, Balleyguier C, Archambaud B, Duffaud F; French Sarcoma Group. Doxorubicin-Trabectedin with Trabectedin Maintenance in Leiomyosarcoma. N Engl J Med. 2024 Sep 5;391(9):789-799. doi: 10.1056/NEJMoa2403394. PMID 39231341
- [Derived] Pautier P, Italiano A, Piperno-Neumann S, Chevreau C, Penel N, Firmin N, Boudou-Rouquette P, Bertucci F, Balleyguier C, Lebrun-Ly V, Ray-Coquard I, Kalbacher E, Bardet A, Bompas E, Collard O, Isambert N, Guillemet C, Rios M, Archambaud B, Duffaud F; French Sarcoma Group. Doxorubicin alone versus doxorubicin with trabectedin followed by trabectedin alone as first-line therapy for metastatic or unresectable leiomyosarcoma (LMS-04): a randomised, multicentre, open-label phase 3 trial. Lancet Oncol. 2022 Aug;23(8):1044-1054. doi: 10.1016/S1470-2045(22)00380-1. Epub 2022 Jul 11. PMID 35835135
- [Derived] Hanvic B, Ray-Coquard I. Gynecological sarcomas: literature review of 2020. Curr Opin Oncol. 2021 Jul 1;33(4):345-350. doi: 10.1097/CCO.0000000000000753. PMID 34009140